CLINICAL TRIAL: NCT03286036
Title: Clinical and Molecular Staging of Lung Cancer Stages I and IIp: Generation and Initial Analysis of a Clinical and Molecular Knowledge Database
Brief Title: Clinical and Molecular Staging of Lung Cancer Stages I and IIp
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Corporacion Parc Tauli (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Consorcio Centro de Investigación Biomédica en Red (CIBER) (Other Government)
Responsible Party: Principal Investigator, Eduard Monsó-Molas, Head of Respiratory Medicine Department, Corporacion Parc Tauli
Other Study IDs: PI12/02040
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Lung Cancer
Keywords: Biomarkers, early detection
MeSH Terms: conditions — Lung Neoplasms | interventions — Biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — tumoral tissue, non-tumoral tissue and blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lung cancer patients: Patients with lung cancer who undergo surgical resection of the tumor
  Interventions: Other: biomarkers

INTERVENTIONS:
Other: biomarkers — This is an observational study, there is no intervention

SUMMARY:
The classification of lung cancer (LC) according to the degree of anatomical extension (TNM) allows the estimation of the prognosis of the patient, although its accuracy is limited. In fact, one third of surgically-treated patients with initial disease have recurrences during follow-up, despite the negativity of node dissection at surgery. The incorporation of genetic, epigenetic and proteomic information to TNM staging will characterize more accurately the lung cancer, and thereby improve the prognostic and the prediction of the therapeutic response in these patients.In this project a prospective cohort of 320 patients with lung cancer staged I-IIp will be studied, combining the clinical and pathologic information available with genetic, epigenetic and proteomic markers in tumour samples, pulmonary tissue, regional nodes and peripheral blood, preserved in suitable systems for the application of complex analytical methodologies. Thus, a knowledge database will be created with the aim of improving the prognostic and prediction capabilities of TNM staging.This project is coordinated with related sub-projects that cover the required laboratory tests on biological samples and with Spanish collaborative group in lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* Able to understand and sign the informed consent

Exclusion Criteria:

* Absence of mediastinal disease

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Lung cancer patients who undergo surgical resection of their tumors in a Spanish hospital with thoracic surgery and pathological anatomy departments
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Cohort creation | 6 years
  Prospective cohort with detailed information of the clinical characteristics at the time of surgery and with biological samples

SECONDARY OUTCOMES:
Biological markers | 3 years
  To identify biological variables with potential prognostic and / or predictive capacity of the therapeutic response, independent of the pathological TNM, in biological samples

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Hospital Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Virgen del Rocio, Seville

IPD SHARING:
Plan to Share IPD: Yes
This is a multicenter study and the patients' samples and clinical data will be available to the study collaborators when the recruitment finishes.

REFERENCES:
- [Background] Monso E, Montuenga LM, Sanchez de Cos J, Villena C; Lung Cancer CIBERES-RTICC-SEPAR-Plataforma Biobanco Pulmonar. Biological Marker Analysis as Part of the CIBERES-RTIC Cancer-SEPAR Strategic Project on Lung Cancer. Arch Bronconeumol. 2015 Sep;51(9):462-7. doi: 10.1016/j.arbres.2014.11.010. Epub 2015 Jan 19. English, Spanish. PMID 25614375